CLINICAL TRIAL: NCT01921439
Title: Matching Brief Smoking Interventions to Stage of Change
Brief Title: OCAST Cessation Study
Acronym: OCAST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma Center for the Advancement of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3262
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Tobacco Smoking Behavior; Cigarette Smoking Behavior; Second Hand Tobacco Smoke; Tobacco Use Cessation
Keywords: smoking; quit smoking; smoking cessation; smoking study; secondhand smoke; smokers
MeSH Terms: conditions — Smoking; Cigarette Smoking; Tobacco Use Cessation; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Feedback (Active Comparator): Participants in this group will receive individualized feedback based on their stage of change. Feedback will include health effects of smoking, money spent per month and per year on cigarettes, time spent smoking compared with time spent doing other daily tasks, and how the participant compares to past study participants in average number of cigarettes per day used and level of addiction.
  Interventions: Behavioral: Personalized Feedback
- No Feedback- Treatment as Usual (TAU) (No Intervention): Participants will take the computer based survey, but will only receive a number to the Oklahoma Tobacco Helpline (Treatment-as-usual condition) instead of feedback.

INTERVENTIONS:
Behavioral: Personalized Feedback — Personalized feedback reflecting the participant's current level of nicotine addiction, money spent on cigarettes, time spent smoking, and health effects of smoking.
  Arms: Feedback

SUMMARY:
The long-term goal is to improve the quality of life of children and their parents who smoke tobacco by facilitating parental smoking cessation in a way that is easy to administer yet effective. We aim to accomplish this goal by administering an interactive computer-based program that will facilitate motivation and readiness to engage in smoking cessation by providing personalized feedback about the financial and health effects of the parent's smoking. We will compare the changes in motivation and readiness to quit smoking after the parent has taken the computer-based program and compare them to the changes in motivation and readiness to quit in parents who receive only information about the Oklahoma Tobacco Helpline. We will also measure salivary cotinine levels in both parents and children, to objectively measure changes in smoking habits and secondhand smoke exposure. Our hypothesis is that our computer-based program will cause a greater increase in motivation and confidence to quit smoking in the group that receives the customized feedback than the group that receives only information about the Tobacco Helpline. We also predict that both parent and child cotinine levels will show a greater decrease in the group randomized to receive personalized feedback.

ELIGIBILITY:
Inclusion Criteria:

* Parent or primary caregiver of a child patient at the OU Children's Physicians General Pediatrics clinics
* Current cigarette user
* Able to read study forms and verbally communicate with the study staff in English

Exclusion Criteria:

* Nonsmokers
* Unable to read or speak English well enough to complete the survey and study tasks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Self-Reported Readiness and Motivation to Quit Smoking | Baseline, 1-month, 6-months, 12-months
  We will assess changes in self-reported readiness and motivation to quit smoking.
Parent and Child Salivary Cotinine | Baseline, 1-month, 6-months, and 12-months
  We will assess change in parent and child salivary cotinine throughout the course of the study.
Change in self-reported cigarette use | baseline, 1-month, 6-months, and 12-months
  We will assess changes in self-reported cigarette use throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Gillaspy, Ph.D., Principal Investigator — The University of Oklahoma Health Sciences Center
Locations (1):
- Oklahoma Tobacco Research Center, Oklahoma City, Oklahoma, United States